CLINICAL TRIAL: NCT01897545
Title: The Role of Renal Denervation in Improving Outcomes of Catheter Ablation in Patients With Atrial Fibrillation and Arterial Hypertension
Brief Title: Combined Treatment of Arterial Hypertension and Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDAFA-030
Record Dates: First submitted 2013-07-03; First posted 2013-07-12 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Arterial Hypertension; Atrial Fibrillation
Keywords: Arterial hypertension; Atrial Fibrillation; Percutaneous renal denervation
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PV isolation (Active Comparator)
  Interventions: Procedure: Circumferential PV isolation
- PV isolation+renal denervation (Active Comparator)
  Interventions: Procedure: PV isolation+renal denervation

INTERVENTIONS:
Procedure: Circumferential PV isolation — The left atrium (LA) and pulmonary veins (PVs) are explored through a transeptal approach. Real-time 3D LA maps are reconstructed by using a nonfluoroscopic navigation system. The ipsilateral left and right PVs are encircled in one lesion line by circumferential PV isolation. Radiofrequency energy is delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and is reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation speed of 17 mL/min. Each lesion is ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 s. The endpoint of circumferential PV isolation is PV isolation. Additional ablation lines are created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the roof of the LA between the two superior PVs. After the end of the procedure the implantable loop recorder is implanted in the parasternal area of the chest.
  Arms: PV isolation
Procedure: PV isolation+renal denervation — The procedure of AF ablation is the same like in the circumferential PV isolation.
  After AF ablation procedure, the angiogram of both renal arteries is performed via femoral access. After that the treatment catheter is introduced into each renal artery and is applied discrete, radiofrequency ablations lasting up to 2 min each and of 8 watts or less to obtain up to six ablations separated both longitudinally and rotationally within each renal artery. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm. After the procedure the control arterial angiogram should be done.
  Arms: PV isolation+renal denervation

SUMMARY:
The purpose of this study is the comparative evaluation of systolic blood pressure (SBP) lowering, atrial fibrillation (AF) recurrence and clinical data in patients with paroxysmal/persistent AF and resistant/non-resistant hypertension, undergoing AF ablation alone or combined with percutaneous renal denervation.

DETAILED DESCRIPTION:
On the basis of the eligibility criteria, patients is assigned by the enrolling physician to one of two strata. The first stratum includes patients with moderate drug-resistant hypertension, defined by the Joint National Committee VII and ESH/ESC guidelines as office BP ≥ 140/90 mm Hg and <160/100 mm Hg. The second stratum includes patients with drug-resistant hypertension, defined by office BP ≥ 160/100 mm Hg.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic drug-refractory AF (with history of failure of ≥2 class I or III antiarrhythmic drugs) in patients referred for catheter ablation of AF
* PAF with ≥1 monthly episodes or PersAF in patients who had already undergone ≥3 electrical cardioversions. PAF was defined as episodes lasting less than 7 days with spontaneous termination. PersAF was defined as lasting more than 7 days before being terminated pharmacologically or by electrical cardioversion.
* Office-based systolic blood pressure of ≥140/90 mm Hg, despite treatment with 3 antihypertensive drugs (including 1 diuretic)
* A glomerular filtration rate ≥45 mL/min/1⋅73 m2, with modification of diet using a renal disease formula

Exclusion Criteria:

* Secondary causes of hypertension
* Severe renal artery stenosis or dual renal arteries
* Congestive heart failure with NYHA II-IV symptoms
* Left ventricular ejection fraction <35%
* Transverse left atrial diameter > 60 mm on transthoracic echocardiography

  1. Previous AF ablation procedure
  2. Treatment with amiodarone
* Previous renal artery stenting or angioplasty
* Type 1 diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
recurrence of > 30 secs of atrial tachyarrhythmia, including AF and left atrial flutter/tachycardia, after a single ablation procedure on no antiarrhythmic drug | 1 year

SECONDARY OUTCOMES:
office blood pressure | 1 year
safety data before and at 3, 6, 9, and 12 months after procedure | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- The Valley Health System, New York, New York, United States
- Athens Euroclinic, Athens, Greece
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Pokushalov E, Romanov A, Katritsis DG, Artyomenko S, Bayramova S, Losik D, Baranova V, Karaskov A, Steinberg JS. Renal denervation for improving outcomes of catheter ablation in patients with atrial fibrillation and hypertension: early experience. Heart Rhythm. 2014 Jul;11(7):1131-8. doi: 10.1016/j.hrthm.2014.03.055. Epub 2014 Mar 29. PMID 24691452